CLINICAL TRIAL: NCT00407771
Title: A Pilot Study of The Effects of a Single High Dose Bolus Tirofiban in Diabetic Patients Undergoing Elective Percutaneous Coronary Intervention
Brief Title: The Effects of Tirofiban in Diabetic Patients Undergoing Elective Percutaneous Coronary Intervention
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jordan Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006-alhaddad
Record Dates: First submitted 2006-12-01; First posted 2006-12-05 (Estimated); Last update posted 2007-10-31 (Estimated); Status verified 2007-10

CONDITIONS: Coronary Artery Disease
Keywords: platelet function assay; Glycoprotein inhibitors; percutaneous coronary intervention; Diabetes Mellitus
MeSH Terms: conditions — Coronary Artery Disease; Diabetes Mellitus | interventions — Tirofiban

INTERVENTIONS:
Drug: Tirofiban

SUMMARY:
* The purpose of this study is to examine the effects of tirofiban on platelet function the Ultegra RPFA in diabetic patients undergoing elective coronary angioplasty and stenting already treated with high loading dose (600mg) clopidogrel.
* About 44 people will be in the study. The study duration is a single hospitalization period during which the angioplasty will be performed in addition to a 30-day post hospitalization follow-up period.
* Patients taking part in the study will be assigned by chance into two groups.

  * Group 1: patients will be treated with the glycoprotein inhibitor, Tirofiban (25mcg/kg over 3 min bolus dose and 0.15 mcg/kg/hr for 12-24 hours), started immediately after insertion of the sheath.
  * Group 2: patients will be treated with equivalent placebo

All patients will be loaded with 600 mg clopidogrel at least 4 hours prior to scheduled intervention.

All patients will have platelet function analyses at baseline and following treatment.

DETAILED DESCRIPTION:
Introduction Diabetes is a major risk factor for coronary artery disease and diabetic patients are considered CAD equivalent in the absence of CAD1. The presence of CAD and diabetes makes the patient at a much higher risk for future morbidity and mortality. Moreover, percutaneous coronary intervention (PCI) in diabetics is associated with a higher risk of major adverse cardiac events (MACE). Several studies have also suggested that the release of cardiac biomarkers during PCI procedures have an independent predictability of a worse prognosis in terms of both morbidity and death. Furthermore, previous investigations suggested that glycoprotein IIb/IIIa inhibitors (GPI) should be used routinely in all diabetics undergoing PCI due to their higher propensity of developing a hyper aggregatory status during such procedures that puts them at a higher risk of developing myocardial injury and subsequent cardiac biomarkers release. However, recent investigation suggested that high dose clopidogrel (600 mg given at least 4 hours prior to intervention) is as protective as Abciximab in low risk patients undergoing elective PCI 2. Thus, high dose clopidogrel preloading without GPI has become the standard for low risk patients undergoing elective PCI. There is limited data in the literature to suggest that routine administration of GPI prior to PCI in diabetic patients with a high dose preloading with clopidogrel is actually beneficial. That is why this trial is being undertaken.

Experience with the high dosage of tirofiban Several studies performed following the completion of TARGET strongly suggested that the 10 µg/kg bolus dose of tirofiban is inadequate3. The TARGET dosing regimen of tirofiban inhibited 20 uMADP-mediated platelet aggregation only by 60-66% from 15-60 minutes after onset of treatment when tested with PPACK as a sample anticoagulant, and as a result of rapid tissue redistribution yielded a tirofiban plasma level of 35-40 ng/mL4. Abciximab, as it was dosed in the TARGET trial, produced a 90-95% inhibition of platelet aggregation in this same time period. This difference in extent of platelet aggregation inhibition was proposed as the reason why more procedure-related ischemic events occurred among subjects receiving tirofiban in the TARGET trial.

To date, several published trials have been described using the single high-dose bolus (SHDB) of tirofiban in various clinical settings. Taken together, more than 600 patients received the SHDB of tirofiban in these clinical trials without evidence of a greater than expected increase in the frequency of bleeding events or thrombocytopenia. A variety of clinical, angiographic, and echocardiographic endpoints all consistently demonstrate that the SHDB of tirofiban is superior to placebo and appears to be comparable to abciximab.

Two trials up to now demonstrated that in the same dosing paradigm SHDB of tirofiban achieves comparable levels of platelet inhibition as does abciximab for patients undergoing PCI4, 5.

The largest experience published by Danzi and colleagues was a 554- patient observational study comparing the safety and efficacy of SHDB tirofiban in PCI patients to a cohort of PCI patients who received abciximab6. Patients were enrolled sequentially: the first 280 received abciximab and the subsequent 274 received HDB tirofiban. The incidence of major bleeding events or access site bleeding complications for patients treated with SHDB tirofiban was less than that seen with abciximab. Moreover, the point estimate of the incidence of in-hospital and 30-day major adverse cardiovascular events (MACE) in the SHDB tirofiban group was actually below that in the abciximab group (5.6% vs. 7.1%; P=0.65). This clinical experience suggests that SHDB tirofiban, administered at the time of PCI, is safe and can produce results similar to abciximab.

Danzi and colleagues published a second clinical trial comparing echocardiographic, angiographic and clinical outcomes in 100 patients with ST-segment elevation myocardial infarction (STEMI) who were treated with SHDB tirofiban versus abciximab7. There was slightly greater improvement in echocardiographic outcomes in patients treated with HDB tirofiban compared with abciximab. Angiographic and clinical outcomes were similar for the two groups. Again, while there was no incidence of major bleeding or severe thrombocytopenia reported for either treatment group, there were actually less episodes of minor bleeding in patients treated with SHDB tirofiban compared with abciximab (4% vs. 8%; P = 0.71). In short, this clinical experience demonstrated that SHDB tirofiban, administered at the time of PCI, was comparable to abciximab in treating STEMI patients undergoing PCI.

A second STEMI manuscript described the study design and demographics of the STRATEGY trial which evaluated STEMI patients who were randomized to receive either SHDB tirofiban + sirolimus eluting stent or abciximab + bare metal stent. This study confirmed the findings of Danzi and co-workers, and also found that the SHBD tirofiban resulted in the same results, as compared to patients treated with Abciximab, with a trend towards a lower bleeding rate with the SHBD tirofiban regimen8 The ADVANCE trial evaluated the efficacy and safety of SHDB tirofiban compared with placebo in treating high-risk patients9. The study enrolled 202 patients with either a single coronary artery occlusion/diabetes, diagnosed NSTEMI, or multivessel coronary artery disease. This trial demonstrated a statistically significant decrease in 6-month MACE or bailout GP IIb/IIIa inhibitor use for patients treated with HDB tirofiban versus placebo (19.8% vs, 34.7%; P=0.01). SHDB tirofiban was shown to significantly reduce the increase in cardiac markers (both troponin I and CK-MB) associated with ischemic events. Subgroup analysis showed a statistically significant decrease in lowering the primary endpoint for diabetic and ACS patients treated with SHDB tirofiban. Finally, there was no major bleeding, need for red blood cell transfusion, or severe thrombocytopenia, and there was no significant difference in even minor bleeding rates between SHDB tirofiban-treated patients and those treated with placebo (4% vs. 1%; P = 0.19).

In summary, these trials represent a significant clinical experience demonstrating the safety and efficacy of the SHDB of tirofiban administered at the time of PCI.

Mechanistic/Pharmacological rationale of benefit expected The use of Tirofiban, given at single high dose bolus, is expected to act on the final common pathway of platelet activation, thus it will completely bypass the COX-1 mediated signal activation (the intracellular pathway on which Aspirin-mediated platelet inhibition is based on). The use of SHDB Tirofiban will result in a dramatic inhibition of platelet activation compared to patients treated with aspirin and clopidogrel alone, determining a significant and profound increase in platelet function which is in contrast to the TACTICS dose10.

Objective of the investigation The Ultegra RPFA is an automated turbidimetric whole blood assay designed to assess platelet function on the basis of the ability of activated platelets to bind to fibrinogen12. The Ultegra RPFA is as accurate and precise as conventional turbidimetric platelet aggregometry13, and a recent study has demonstrated that the measurements are not operator dependent or influenced by concomitant medications, hematologic parameters, or demographics14.

The objectives of this proposal is to conduct a pilot study examining the platelet function using the Ultegra RPFA in diabetic patients undergoing elective PCI when treated with tirofiban and high loading dose (600mg) clopidogrel versus high loading dose clopidogrel alone.

Additional assays of flow cytometry and platelet monocyte aggregation will be analyzed in a similar fashion before and after treatment.

Baseline blood samples will also be assessed for lipid profile, Hs-CRP, FBS, renal function, liver function, CBC and HbA1c.

Null Hypothesis It is expected that tirofiban arm will provide over 90% platelet aggregation inhibition compared to the Clopidogrel alone arm which will provide a maximum of 50% platelet aggregation inhibition. Therefore, an expected difference of 40% in platelet inhibition is anticipated in this pilot trial.

End points

The primary endpoint:

To investigate the magnitude of platelet aggregation inhibition using SHBD tirofiban with clopidogrel versus clopidogrel alone before randomization, 10 minutes (t=0) and 8 hours (t=8) post tirofiban administration.

Observational point:

1. The difference of flow cytometry and platelet monocyte aggregation between the two groups.
2. The incidence of troponin T release 12 hours post PCI among the two groups.
3. The difference in mean troponin T between the groups at 12 hours post PCI.
4. Major adverse cardiac events (MACE) at 24 hours and 30 days post PCI.

Follow-up All patients screened (independent of their AR status) will be clinically followed-up for 1 month to evaluate observational point.

Study Design and Procedures:

Type of study This is a randomized, open label, placebo controlled (with bailout tirofiban as rescue) single center study.

Statistical Considerations

Number of patients The study enrollment will be stopped as soon as a total of 44 patients randomized to receive Tirofiban (in addition to Aspirin, Heparin and 600mg Clopidogrel) vs. Aspirin, Heparin and 600mg clopidogrel alone and who actually undergo PCI.

Statistical Analysis Two analyses will be performed; the first is based on intention to treat and the other considering bailout tirofiban administration and will reflect actual treatment. Since the primary outcomes are related to operator independent analysis of platelet function, we do not expect bias in the interpretation of final results and conclusions.

Main Study Flow 44 Diabetic patients referred for elective PCI will be randomized into two groups. Group 1: patients will be treated with the GPI, Tirofiban (25mcg/kg over 3 min bolus dose and 0.15 mcg/kg/hr for 12-24 hours), started immediately after insertion of the sheath. Group 2: patients will be treated with equivalent placebo.

All patients will be loaded with 600 mg clopidogrel at least 4 hours prior to scheduled intervention.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients with coronary artery disease undergoing elective percutaneous coronary intervention

Exclusion Criteria:

* Ongoing ST-segment elevation myocardial infarction (MI)
* Administration of abciximab during the previous two weeks
* Serum creatinine more than 2.5 mg/dl (221 micro-mol/L)
* Ongoing bleeding or bleeding diathesis
* Previous stroke in the last six months
* Major surgery within the previous six weeks
* Platelet count <100.000 per cubic mm
* Subjects who received low-molecular-weight heparin, tirofiban, or eptifibatide within the 10 hours prior to randomization
* Subjects on oral anticoagulation medication (coumarin derivatives) within the last 7 days unless PT-INR <1.5 times the control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2007-11; Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
The magnitude of platelet aggregation inhibition before randomization, 10 minutes (t=0) and 8 hours (t=8) post tirofiban administration using the Ultegra RPFA assay.

SECONDARY OUTCOMES:
The difference of flow cytometry and platelet monocyte aggregation between the two groups.
The incidence of troponin T release 12 hours post PCI among the two groups.
The difference in mean troponin T between the groups at 12 hours post PCI.
Major adverse cardiac events (MACE) at 24 hours and 30 days post PCI.

CONTACTS AND LOCATIONS:
Overall Officials: Imad A Alhaddad, MD, Principal Investigator — Jordan Cardiovascular Center
Locations (1):
- Jordan Hospital, Amman, Jordan

REFERENCES:
- [Background] Danzi GB, Capuano C, Sesana M, Baglini R. Preliminary experience with a high bolus dose of tirofiban during percutaneous coronary intervention. Curr Med Res Opin. 2003;19(1):28-33. doi: 10.1185/030079902125001380. PMID 12661777
- [Background] Schneider DJ, Herrmann HC, Lakkis N, Aguirre F, Wan Y, Aggarwal A, Kabbani SS, DiBattiste PM. Enhanced early inhibition of platelet aggregation with an increased bolus of tirofiban. Am J Cardiol. 2002 Dec 15;90(12):1421-3. doi: 10.1016/s0002-9149(02)02892-8. No abstract available. PMID 12480064
- [Background] Valgimigli M, Percoco G, Barbieri D, Ferrari F, Guardigli G, Parrinello G, Soukhomovskaia O, Ferrari R. The additive value of tirofiban administered with the high-dose bolus in the prevention of ischemic complications during high-risk coronary angioplasty: the ADVANCE Trial. J Am Coll Cardiol. 2004 Jul 7;44(1):14-9. doi: 10.1016/j.jacc.2004.03.042. PMID 15234398
- [Background] Kimmelstiel C, Badar J, Covic L, Waxman S, Weintraub A, Jacques S, Kuliopulos A. Pharmacodynamics and pharmacokinetics of the platelet GPIIb/IIIa inhibitor tirofiban in patients undergoing percutaneous coronary intervention: implications for adjustment of tirofiban and clopidogrel dosage. Thromb Res. 2005;116(1):55-66. doi: 10.1016/j.thromres.2004.11.011. Epub 2004 Dec 8. PMID 15850609
- [Background] Bonz AW, Lengenfelder B, Strotmann J, Held S, Turschner O, Harre K, Wacker C, Waller C, Kochsiek N, Meesmann M, Neyses L, Schanzenbacher P, Ertl G, Voelker W. Effect of additional temporary glycoprotein IIb/IIIa receptor inhibition on troponin release in elective percutaneous coronary interventions after pretreatment with aspirin and clopidogrel (TOPSTAR trial). J Am Coll Cardiol. 2002 Aug 21;40(4):662-8. doi: 10.1016/s0735-1097(02)02014-4. PMID 12204495
- [Background] Wheeler GL, Braden GA, Steinhubl SR, Kereiakes DJ, Kottke-Marchant K, Michelson AD, Furman MI, Mueller MN, Moliterno DJ, Sane DC. The Ultegra rapid platelet-function assay: comparison to standard platelet function assays in patients undergoing percutaneous coronary intervention with abciximab therapy. Am Heart J. 2002 Apr;143(4):602-11. doi: 10.1067/mhj.2002.121734. PMID 11923796
- [Background] Gurbel PA, Bliden KP, Zaman KA, Yoho JA, Hayes KM, Tantry US. Clopidogrel loading with eptifibatide to arrest the reactivity of platelets: results of the Clopidogrel Loading With Eptifibatide to Arrest the Reactivity of Platelets (CLEAR PLATELETS) study. Circulation. 2005 Mar 8;111(9):1153-9. doi: 10.1161/01.CIR.0000157138.02645.11. Epub 2005 Feb 28. PMID 15738352